CLINICAL TRIAL: NCT02534649
Title: Bergonie Institut Profiling : Fighting Cancer by Matching Molecular Alterations and Drugs in Early Phase Trials
Acronym: BIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB2015-09
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor; Hematological Malignancy
Keywords: Molecular profiling; Genomic alteration; Advanced cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Other): Newly obtained biopsy and Blood samples collection
  Interventions: Procedure: Newly obtained biopsy and Blood samples collection

INTERVENTIONS:
Procedure: Newly obtained biopsy and Blood samples collection — For each patient:
  * Frozen and paraffin embedded tumor material (archival or new biopsy) will be obtained for genetic profiling
  * Four blood samples will be obtained for genetic profiling and assessment of markers The results of each tumor profile will be discussed within a multidisciplinary tumor board which aims at discussing the genomic profiles and at providing a therapeutic decision for each patient.
  Patients for whom no molecular aberration has been identified will be treated at the discretion of the investigator and followed until death or study termination whichever occurs first.
  All the patients carrying a molecular aberration will be proposed to enter in a clinical trial depending on the possibility of inclusion at the time of molecular report.

SUMMARY:
This is a biology driven, monocentric study designed to identify actionable molecular alterations in cancer patients with advanced disease.

In this trial, high throughput analysis will be carried out using next generation sequencing, and immunological profiling.

Patients included in the BIP study and for whom a targetable genomic alteration had been identified might be subsequently included in an early phase trials running at Institut Bergonie or another French hospital.

DETAILED DESCRIPTION:
The need to 'personalize' cancer therapy has been recognized, with specific biomarkers which will be used to direct targeted agents only to those patients deemed most likely to respond. This "personalized cancer medicine" requires two critical steps: first, a comprehensive assessment of the biological characteristics of tumors from each individual, and second, validated biomarkers to identify the subgroups of patients who are most likely to benefit from a given therapy and the next-generation sequencing provides unprecedented opportunities to draw a comprehensive picture of genetic aberrations involve in immunotherapy sensitivity and ultimately enable individualized treatment.

The main objective of this study is to use next generation sequencing technologies to identify actionable molecular alterations in cancer patients with advanced disease included in the study. This study will provide a fully integrated view of the molecular profile of the tumor for each patient included in the study. Such tumor profile will be used by clinicians to tailor therapies of patients in specific early phase clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Histology: solid malignant tumor or hematological malignancy,
3. Deleted MSA9
4. Deleted MSA9,
5. Deleted MSA9,
6. Deleted MSA9,
7. Patient with a social security in compliance with the French law relating to biomedical research (Article L.1121-11 of French Public Health Code),
8. Voluntary signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

1. Deleted MSA9
2. Deleted MSA9
3. Deleted MSA9
4. Deleted MSA9
5. Deleted MSA9
6. Deleted MSA9
7. Deleted MSA9
8. Deleted MSA9
9. Individuals deprived of liberty or placed under guardianship
10. Pregnant or breast feeding women,
11. Previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients presenting at least one genomic alteration | 1 month
  The proportion of patients with advanced cancer presenting at least one genomic alteration will be described in the NGS population and reported using the proportion. The 95% two-sided confidence limits (95%CI) will be provided for the calculated rate (binomial law).

SECONDARY OUTCOMES:
- Utilization rates of molecular profiling information (including utilization of information for standard regimens or clinical trials of molecularly targeted therapies) | Utilization rates of molecular profiling information will be evaluated until the date of death from any cause, assessed up to 36 months
  Utilization rates of molecular profiling information (including utilization of information for standard regimens or clinical trials of molecularly targeted therapies. For a patient with NGS results available, utilization of molecular profiling information is defined as :
  * Inclusion in a clinical trial assessing a drug matched with the genetic profile
  * Treatment with an approved drug matched with the genetic profile
Rate of molecular screening failure | Molecular screening failure will be assessed at 1 month
  Rate of molecular screening failure. Molecular screening failure is defined as the impossibility to provide genetic profiling because as a result of inadequate tissue or DNA quantity or quality.
Safety of biopsies procedures (when applicable) graded according to NCI-CTC v4.0. | Safety will be assessed 1 month after biopsy
  Safety of biopsies procedures (when applicable) graded according to NCI-CTC v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ITALIANO, MD, PhD, Study Chair — Institut Bergonié
Locations (7):
- France (7):
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Clinique Tivoli-Ducos, Bordeaux
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Hospitalier de Pau, Pau
  - Clinique Marzet, Pau
  - Centre Eugène Marquis, Rennes

REFERENCES:
- [Derived] Guegan JP, Peyraud F, Dadone-Montaudie B, Teyssonneau D, Palmieri LJ, Clot E, Cousin S, Roubaud G, Cabart M, Leroy L, Lebreton C, Rey C, Lara O, Odin O, Brunet M, Vanhersecke L, Gruyters EO, Achour I, Belcaid L, Le Moulec S, Grellety T, Bessede A, Italiano A. Analysis of PD1, LAG3, TIGIT, and TIM3 expression in human lung adenocarcinoma reveals a 25-gene signature predicting immunotherapy response. Cell Rep Med. 2024 Dec 17;5(12):101831. doi: 10.1016/j.xcrm.2024.101831. Epub 2024 Nov 25. PMID 39591972